CLINICAL TRIAL: NCT02836080
Title: Integrated Collaborative Care Teams to Enhance Service Delivery to Youth With Mental Health and Substance Use Challenges: Protocol for a Pragmatic Randomized-controlled Trial
Brief Title: Integrated Collaborative Care Teams for Youth With Mental Health and/or Addiction Challenges (YouthCan IMPACT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: East Metro Youth Services (Other); Delisle Youth Services (Unknown); LOFT Community Services (Other); The Sashbear Foundation (Unknown); The Anne Johnston Health Station (Unknown); South East Toronto Family Health Team (Unknown); Institute for Clinical Evaluative Sciences (Other); Medical Psychiatry Alliance (Other); Graham Boeckh Foundation (Other); The Ontario Spor Support Unit (Other)
Responsible Party: Principal Investigator, Joanna Henderson, Director, Margaret and Wallace McCain Centre for Child, Youth and Family Mental Health; Associate Professor of Psychiatry, University of Toronto, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #012/2016
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Mental Disorders; Addiction
Keywords: Mental Health; Randomized; Pragmatic; Integrated Collaborative Care; Addiction; Youth
MeSH Terms: conditions — Mental Disorders; Behavior, Addictive; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated Collaborative Care Team (Experimental): Integrated Collaborative Care Team (ICCTs) are housed in the local community to improve youth access, in three neighborhoods across Toronto (East Metro Youth Services [EMYS]-Scarborough, EMYS-Southeast Toronto, and Delisle Youth Services-Central Toronto). Each ICCT will include a variety of service providers and coordinated patient care delivering evidence-informed interventions in a stepped-care model.
  Interventions: Behavioral: Integrated Collaborative Care Team (ICCT)
- Treatment as Usual (TAU) (Active Comparator): The comparator arm consists of out-patient TAU in a hospital setting and will occur at one of four outpatient hospital sites across Toronto.
  Partners include the following four hospitals: Hospital for Sick Children (SickKids), the Centre for Addiction and Mental Health (CAMH), Michael Garron Hospital (formerly the Toronto East General Hospital), and Sunnybrook Hospital.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Integrated Collaborative Care Team (ICCT) — An integrated, collaborative pathway of needs-based services. ICCTs will offer a wide variety of services, including Solution-Focused Brief Therapy (SFBT) on a scheduled and walk-in basis, care navigators, various clinician-guided interventions, psychiatry, nurse practitioner services, access to primary care, and peer support, all co-located in youth-friendly, community-based clinics. For each intervention, standardized intervention protocols will be used.
  Arms: Integrated Collaborative Care Team
Other: Treatment as Usual (TAU) — Standard out-patient treatment provided at each participating hospital site. This typically entails referral to a psychiatrist at the participating hospital, who will provide assessment and treatment, with referral to appropriate services, guided by local treatment protocols.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Among youth, the prevalence of mental health and addiction (MHA) disorders is roughly 20%, yet youth are challenged to access services in a timely fashion. To address MHA system gaps, this study will test the benefits of an Integrated Collaborative Care Team (ICCT) model for at-risk youth with MHA challenges. In partnership with community agencies, adolescent psychiatry hospital departments, and family health teams, investigators have developed an innovative model of service provision involving rapid access to MHA services. This model will be implemented and compared to the usual treatment youth receive in hospital-based, outpatient, mental health clinics in Toronto. A rapid, systematic, approach to MHA services geared to need in a youth-friendly environment is expected to result in better MHA outcomes for youth. Moreover, the ICCT approach is expected to decrease service wait-times, be more youth- and family-centred, and be more cost-effective.

DETAILED DESCRIPTION:
This study is a pragmatic randomized control trial (RCT) with random allocation occurring within each hospital site to either treatment as usual (TAU) (4 out-patient hospital sites) or treatment at one of 3 community-based Integrated Collaborative Care Teams (ICCTs). A total of 500 youth aged 14-18 with mental health and/or addictions (MHA) concerns, referred for out-patient services at one of four local hospitals, will be randomized to receive ICCT care versus TAU. For each youth, a primary caregiver will also be recruited into the study, if available.

With wide inclusion criteria and a design meant to emulate a "real world" setting, this study will rigorously evaluate a service delivery model composed of multiple interventions for youth presenting with a broad range of MHA problems. The ICCT is expected to result in better MHA outcomes, show better performance indicators, and be more cost-effective than TAU.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Aged 14 - 17 years 11 months
3. New referrals to one of the four participating hospitals for out-patient MHA services
4. Among the population regularly accepted for out-patient services at that hospital

Exclusion Criteria:

1. Referral for specialty forensic or firesetting treatment
2. Moderate to severe intellectual disability or autism without MHA problems
3. Primary diagnosis of an eating disorder
4. Active psychosis or imminent risk of self-harm requiring immediate intervention
5. Inability to read and write English or to consent to the study

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 247 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Youth functioning | One year
  Measured using the Columbia Impairment Scale (CIS)

SECONDARY OUTCOMES:
Clinical improvement | One year
  Measured using Strengths and Difficulties Questionnaire
Problematic substance use | One year
  Assessed using the GAIN Short Screener and the substance use table of the Adolescent Alcohol and Drug Involvement Scale
Satisfaction with the service models | One year
  Assessed using the Ontario Perception of Care Tool for Mental Health and Addictions
Continuity of care | One year
  Measured using the Continuity of Care in Children's Mental Health questionnaire
Goal attainment | One year
  Measured using a custom form indicating goals established by the youth and caregiver at intake, followed by a rating of goal attainment
Client empowerment and engagement | One year
  Measured using the Family Empowerment Scale for caregivers, and the Youth Efficacy/Empowerment Scale for youth
Caregiver burden | One year
  Measured using the Burden Assessment Scale
Quality-adjusted life years (QALYs) | One year
  Measured using the Assessment of Quality of Life-6D (AQOL-6D)
Cost-effective analysis (CEA) and a cost-utility analysis (CUA) | One year
  Incremental costs of ICCT compared to TAU (treatment as usual) in improving health outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Henderson, Ph.D., C.Psych, Principal Investigator — Director, Margaret and Wallace McCain Centre for Child, Youth and Family Mental Health; Clinician Scientist, Centre for Addiction and Mental Health; Associate Professor, Dept. of Psychiatry, University of Toronto; Peter Szatmari, MD, FRCPC, Principal Investigator — Chief, Child and Youth Mental Health Collaborative, The Hospital for Sick Children and Centre for Addiction and Mental Health; Professor and Head of the Division of Child and Youth Mental Health, University of Toronto; Amy Cheung, MD, FRCPC, Principal Investigator — Associate Scientist, Evaluative Clinical Sciences, Hurvitz Brain Sciences Research Program, Sunnybrook Research Institute; Associate Professor, Department of Psychiatry, University of Toronto; Kristin Cleverley, RN, Ph.D., Principal Investigator — CAMH Chair in Mental Health Nursing Research; Assistant Professor, University of Toronto; Clinician-Scientist, Margaret and Wallace McCain Centre for Child, Youth & Family Mental Health, Centre for Addiction and Mental Health; Gloria Chaim, M.S.W., Principal Investigator — Associate Director, Child Youth and Family Services; Head, Community Engagement and Partnership, Margaret and Wallace McCain Centre for Child, Youth and Family Mental Health, CAMH; Assistant Professor, Dept. of Psychiatry, University of Toronto
Locations (5):
- Canada (5):
  - North York General Hospital, Toronto, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Quinlan-Davidson M, Henderson JL, Szatmari P, Cheung A, Dixon M, Relihan J, Singer D, Hawke LD, Cleverley K. A qualitative study exploring youth's experiences of hospital- and integrated community-based mental health services: the YouthCan IMPACT initiative. BMC Psychiatry. 2025 Nov 12;25(1):1084. doi: 10.1186/s12888-025-07523-7. PMID 41225406
- [Derived] Henderson J, Szatmari P, Cleverley K, Ma C, Hawke LD, Cheung A, Relihan J, Dixon M, Quinlan-Davidson M, Moretti M, de Oliveira C, Lee A, Courtney DB, O'Brien D, McDonald H, Lemke K, Pignatiello T, Monga S, Kozloff N, Solomon L, Andrade BF, Barwick M, Charach A, Courey L, Darnay K, Kurdyak P, Lin E, Shan D. Integrated Collaborative Care for Youths With Mental Health and Substance Use Challenges: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e259565. doi: 10.1001/jamanetworkopen.2025.9565. PMID 40358950
- [Derived] Krause KR, Lee A, Shan D, Cost KT, Hawke LD, Cheung AH, Cleverley K, de Oliveira C, Quinlan-Davidson M, Moretti ME, Henderson JL, Ma C, Szatmari P. Minimally important change on the Columbia Impairment Scale and Strengths and Difficulties Questionnaire in youths seeking mental healthcare. BMJ Ment Health. 2025 Jan 22;28(1):e301425. doi: 10.1136/bmjment-2024-301425. PMID 39848629
- [Derived] Henderson JL, Cheung A, Cleverley K, Chaim G, Moretti ME, de Oliveira C, Hawke LD, Willan AR, O'Brien D, Heffernan O, Herzog T, Courey L, McDonald H, Grant E, Szatmari P. Integrated collaborative care teams to enhance service delivery to youth with mental health and substance use challenges: protocol for a pragmatic randomised controlled trial. BMJ Open. 2017 Feb 6;7(2):e014080. doi: 10.1136/bmjopen-2016-014080. PMID 28167747
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital — http://www.camh.net/research